CLINICAL TRIAL: NCT03486613
Title: Patient-reported Outcome Measures Collected in DANBIO Reported Via a Smartphone App Versus a Touch Screen Solution in an Outpatient Clinic Among Patients With Inflammatory Arthritis: A Randomised Cross-over Agreement Study
Brief Title: PROM Collected Via a Smartphone App Versus a Touch Screen Solution Among Patients With Inflammatory Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Salome Kristensen (Other)
Responsible Party: Sponsor-Investigator, Salome Kristensen, MD, PhD, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2018-000367
Record Dates: First submitted 2018-02-08; First posted 2018-04-03 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Rheumatoid Arthritis; Psoriatic Arthritis; Axial Spondyloarthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic; Axial Spondyloarthritis

STUDY DESIGN:
Intervention Model Description: A randomised, within-participants, open, cross-over design trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group AT (Other): PROM registration via the DANBIO App on a smartphone and thereafter the touch screen solution
  Interventions: Other: PROM registration via the DANBIO App on a smartphone; Other: PROM registration via the touch screen solution
- Group TA (Other): PROM registration via the touch screen solution and thereafter the DANBIO App
  Interventions: Other: PROM registration via the DANBIO App on a smartphone; Other: PROM registration via the touch screen solution

INTERVENTIONS:
Other: PROM registration via the DANBIO App on a smartphone — PROM data is reported through the DANBIO smartphone app
Other: PROM registration via the touch screen solution — PROM data is reported through the touch screen solution

SUMMARY:
A randomised, within-participants cross-over design trial including 60 patients with rheumatoid arthritis, psoriatic arthritis and axial spondyloarthritis. The participants will be randomised to data registration of patient reported outcome measures (PROM) through the DANBIO app on a smartphone first and thereafter via the touch screen solution at the rheumatology outpatient clinic or vice versa. Outcomes are the following PROM: HAQ, VAS pain, VAS fatigue, VAS global Health, BASDAI, BASFI, PASS, Anchoring question, DAS28crp and ASDAS.

DETAILED DESCRIPTION:
The study is a randomised, within-participants cross-over design trial including 60 patients with rheumatoid arthritis (RA) (20), psoriatic arthritis (PsA) (20) and axial spondyloarthritis (SpA) (20) from the Rheumatology outpatient clinic at Aalborg University Hospital. The participants will be randomised in ratio 1:1 to:

* Group AT (App → Touch) (30 participants) the participant reports data through the DANBIO app on a smartphone first and after a "washout period" of one day via the touch screen solution at the rheumatology outpatient clinic.
* Group TA (Touch → App) (30 participants): the participant reports data through the touch screen solution at the rheumatology outpatient clinic and after a "washout period" of one day via the DANBIO app on a smartphone.

The primary objective is to evaluate whether electronic reporting of PROM through the DANBIO smartphone app is comparable to the traditional touch screen solution in the rheumatology outpatient clinic among patients with inflammatory arthritis in standard clinical care. The primary outcome is HAQ. Secondary outcomes are: VAS pain, VAS fatigue, VAS global Health, BASDAI, BASFI, PASS, Anchoring question, DAS28crp and ASDAS. DAS28crp are estimated using a fixed level for C-reactive protein (CRP) level of 6, swollen joint count of 0.5 and tender joint count of 1. ASDAS are estimated using a fixed level for CRP of 6. These data are based on DANBIO registrations of patients with RA, PsA or SpA from the rheumatology outpatient clinic at Aalborg University Hospital. DAS28crp and ASDAS are estimated from the PROM data to give the clinician an overview of PROM correlating to e.g. remission or high disease activity.

ELIGIBILITY:
Inclusion Criteria:

A participant will be eligible for study participation if he/she meets the following criteria:

* Diagnosed in DANBIO with RA, PsA or SpA
* Is currently treated and monitored at the rheumatology outpatient clinic at Aalborg University Hospital
* Have previously reported PROM in DANBIO through the touch screen solution at the rheumatology outpatient clinic ≥ 3 times

Exclusion Criteria:

A participant cannot be included in the study if he/she meets any of the following criteria:

* Inability to provide informed consent or unwilling to comply with the study protocol
* Diagnosis of RA, PsA or SpA ≤ 12 months
* Does not have access to a smartphone that can download and run the DANBIO app
* Not able to understand written Danish i.e. cannot understand the Danish version of the PROM questionnaires
* Reduced sight in such degree that the participant cannot read the questionnaire in the smartphone app/on the touch-screen with e.g. glasses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-04-24 (Actual); Primary Completion 2019-09-12 (Actual); Study Completion 2019-09-12 (Actual)

PRIMARY OUTCOMES:
Change in Health Assessment Questionnaire (HAQ) | day 1 (first data registration) and day 3 (second data registration)
  Assess the patient's physical function

SECONDARY OUTCOMES:
Visual Analogue Scale for Pain | day 1 (first data registration) and day 3 (second data registration)
  The patient's assessment of pain on a scale from 0-100 within the last week. The left of the scale (0) signifies the absence of pain and the right end (100) maximum pain.
Visual Analogue Scale for fatigue | day 1 (first data registration) and day 3 (second data registration)
  The patient's assessment of fatigue on a scale from 0-100 within the last week. The left of the scale (0) signifies the absence of fatigue and the right end (100) maximum fatigue.
Patient Global Visual Analogue Scale | day 1 (first data registration) and day 3 (second data registration)
  The patient's global assessment of disease activity (arthritis severity) on a scale from 0-100 within the last week. The left of the scale (0) signifies the absence of arthritis activity and the right end (100) maximum arthritis activity.
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | day 1 (first data registration) and day 3 (second data registration)
  The patient's assessment of essential symptoms in axial arthritis. The questionnaire consist of six questions regarding essential symptoms in axial arthritis answered on a Visual Analogue Scale from 0-100. The left of the scale (0) signifies the absence of symptoms and the right end (100) maximum symptoms. The patient's answer for each individual question are added to a combined score of 0-100, where 0 signifies the absence of symptoms and 100 maximum symptoms.
Bath Ankylosing Spondylitis Functional Index (BASFI) | day 1 (first data registration) and day 3 (second data registration)
  The patient's assesment of physical function. The questionnaire consist of ten questions regarding physical function in axial arthritis answered on a Visual Analogue Scale from 0-100. The left of the scale (0) signifies the absence of physical limitations and the right end (100) maximum physical limitations. The patient's answer for each individual question are added to a combined score of 0-100, where 0 signifies the absence physical limitations and 100 maximum physical limitations.
Patient Acceptable Symptom State (PASS) | day 1 (first data registration) and day 3 (second data registration)
  The patient's assessment of acceptable symptom state. Consist of one question answered with "yes" or "no". The question is: ''Take into account all the ways in which your arthritis has affected you in the past 48 hours. If you were to remain for the next few months as you are today, would it be acceptable to you?"
Anchoring question | day 1 (first data registration) and day 3 (second data registration)
  The patient's assessment of change in arthritis activity since last visit
Disease Activity Score 28 joints C-reactive protein (DAS28crp) | day 1 (first data registration) and day 3 (second data registration)
  Composite score used as a measurement of disease activity in patients with peripheral arthritis. The DAS28crp score is based on 28 joint count for tenderness (TJC28) and swelling (SJC28), Patient Global Visual Analogue Scale (GH) and CRP level (CRP). The DAS28crp equation is: DAS28crp = 0.56square root(TJC28) + 0.28square root(SJC28) + 0.36ln(CRP + 1) + 0.014(GH) + 0.96. ASDAS = 0.12*Back Pain + 0.06*Morning Stiffness + 0.11*Patient Global + 0.07*Peripheral Pain/Swelling + 0.58*Ln(CRP+1)0.96-9.4 where a score under 2.6 is remission, a score between 2.6-3.1 is low disease activity, a score of 3.2-5.1 is moderate disease activity and a score of 5.1 or higher is high disease activity.
Ankylosing Spondylitis Disease Activity Score (ASDAS) | day 1 (first data registration) and day 3 (second data registration)
  Composite score used as a measurement of disease activity in patients with axial arthritis. The ASDAS score is based on some of the questions from the BASDAI questionnaire and C-reative protein (CRP). The ASDAS equation is: ASDAS = 0.12*Back Pain + 0.06*Morning Stiffness + 0.11*Patient Global + 0.07*Peripheral Pain/Swelling + 0.58*Ln(CRP+1). The scale ranges from 0.6 to infinite where a score under 1.3 is remission, a score between 1.3-2.0 is moderate disease activity, a score of 2.1-3.5 is high disease activity and a score of higher than 3.5 is very high disease activity.

CONTACTS AND LOCATIONS:
Overall Officials: Salome Kristensen, MD, PhD, Principal Investigator — Department of Rheumatology, Aalborg University Hospital
Locations (1):
- Department of Rheumatology, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No